CLINICAL TRIAL: NCT05372393
Title: Carpal Tunnel Release Under Local Anaesthesia With or Without Distal Median Nerve Block - a Protocol of a Double Blinded Randomised Controlled Trial
Brief Title: Carpal Tunnel Release Under Local Anaesthesia With or Without Distal Median Nerve Block
Acronym: PERSONNEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUH5203140
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; carpal tunnel release; local anaesthesia; surgery; wide-awake local anaesthesia with no tourniquet; nerve block
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Two concurrent study groups
Who Masked: Participant, Investigator
Masking Description: Masking is double blinded (patient and investigators). The trial patients are blinded to the randomization. They can't see to the operation field. In the local anaesthesia group care provider pinches from the area of median nerve blockade prior to performing local anaesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local infiltration anaesthesia in carpal tunnel release (Active Comparator): The investigators allocate 59 patients in this arm. It serves as the control group, who receives local infiltration anaesthesia.
  Interventions: Procedure: Local infiltration anaesthesia in carpal tunnel release
- Distal median nerve block with local infiltration anaesthesia in carpal tunnel release (Experimental): The investigators allocate 59 patients in this arm. It serves as the experimental group, who receives local infiltration anaesthesia and distal median nerve block.
  Interventions: Procedure: Distal median nerve block with local infiltration anaesthesia in carpal tunnel release

INTERVENTIONS:
Procedure: Local infiltration anaesthesia in carpal tunnel release — The anaesthetic cocktail consists of 1 ml of (7.5%) sodium bicarbonate (Natriumbicarbonate Braun 75mg/ml), 4,5 ml of lidocaine with adrenaline 1% (Lidocain cum adrenalin 10 mg/ml), 4,5 ml of bupivacaine with adrenaline 0.5% (Marcain cum adrenalin 5mg/ml +5 µg/ml). The anaesthetic cocktail must be prepared in the above-mentioned order to avoid possible precipitation. A 24-gauge hypodermic needle and 10 ml syringe are used to inject the solution. The care provider pinches from the area of median nerve blockade prior to performing local anaesthesia. All the anaesthetic solution is injected locally. Additional anaesthetic solution can be injected locally if necessary.
  Arms: Local infiltration anaesthesia in carpal tunnel release
Procedure: Distal median nerve block with local infiltration anaesthesia in carpal tunnel release — The anaesthetic cocktail consists of 1 ml of (7.5%) sodium bicarbonate (Natriumbicarbonate Braun 75mg/ml), 4,5 ml of lidocaine with adrenaline 1% (Lidocain cum adrenalin 10 mg/ml), 4,5 ml of bupivacaine with adrenaline 0.5% (Marcain cum adrenalin 5mg/ml +5 µg/ml). The anaesthetic cocktail must be prepared in the above-mentioned order to avoid possible precipitation. A 24-gauge hypodermic needle and 10 ml syringe are used to inject the solution. Half of the anaesthetic solution is injected into the median nerve area 5-7 cm proximally from the distal wrist crease. The other half is injected locally. Additional anaesthetic solution can be injected locally if necessary.
  Arms: Distal median nerve block with local infiltration anaesthesia in carpal tunnel release

SUMMARY:
Carpal tunnel syndrome (CTS) is the most commonly appearing entrapment neuropathy of the upper extremity. Treatment options include both non-operative and operative methods. Surgical treatment, carpal tunnel release (CTR), involves division of the transverse carpal ligament. Surgery can be performed under axillary or intravenous block, or general anaesthesia. There are no prior randomised controlled trials (RCT) comparing local infiltration anaesthesia to local infiltration anaesthesia augmented with a distal median nerve block in CTR.

The aim of this trial is to investigate whether adding a distal median nerve block to local anaesthesia reduces the patient's perceived pain level for up to 72 hours after CTR, compared to using only local anaesthesia, i.e., an anaesthesia mixture injected solely in and around the planned incision and nerve release. The null hypothesis is that the use of distal median nerve block with local anaesthesia does not reduce pain after CTR compared to pure local anaesthesia.

PERSONNEL (carPal tunnEl ReleaSe lOcal iNfiltratioN mEdian bLockade) is a double-blinded, i.e., patient and investigators, RCT in patients with CTS. Patients will be randomly divided into two parallel trial groups, 1:1 in size to each other. Fifty-nine patients will be needed for each group to have adequate power. The primary outcome is the pain level perceived by the patient after the procedure during the first 72 hours using the Visual Analogue Scale (VAS). Secondary outcomes include patient-rated outcome measures, safety, the entire consumption of pain killers after the surgery during the first 72 hours postoperatively, pain of performing the anaesthesia, and pain during and after the operation.

No trial comparing local anaesthesia to local anaesthesia augmented with distal median nerve block has been published before. There is also no trial noting individual tolerance to pain. The quality of the median nerve block at the wrist has been achieved by using sensory or sensory-motor nerve stimulation and has been proven effective. This increases trust in the effectiveness of the treatment method, but it still needs to be adequately proven which is the goal of this trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* CTS verified by nerve conduction studies
* Symptoms suitable for CTS

Exclusion Criteria:

* Recurrent CTS
* Peripheral neuropathies
* Known allergy to the trial drugs
* Profound cognitive impairment
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The pain level perceived by the patient after the procedure using Visual Analogue Scale (VAS) | Postoperatively during the first 72 hours after the operation
  The investigators measure the pain level perceived by the patient after the procedure every fourth hour while awake until third night postoperatively using VAS. The first assessment is performed four hours after the surgery. The mean VAS is calculated from all time points over the 72-hour period. The Visual analogue Scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable.

SECONDARY OUTCOMES:
Pressure pain (VAS) | Immediately after the infiltration of anaesthetic solution
  The investigators ask the patients to evaluate the pressure pain that the infiltration of the anaesthetic solution caused using Visual Analogue Scale (VAS). The Visual Analogue Scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable.
Burning pain (VAS) | Immediately after the infiltration of anaesthetic solution
  The investigators ask the patients to evaluate the burning pain that the infiltration of the anaesthetic solution caused using Visual Analogue Scale (VAS). The Visual Analogue Scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable.
Needle sting pain (VAS) | Immediately after the infiltration of anaesthetic solution
  The investigators ask the patients to evaluate the needle sting pain that the infiltration of the anaesthetic solution caused using Visual Analogue Scale (VAS). The Visual Analogue Scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable.
Total pain during the injection of the anaesthetic solution (VAS) | Immediately after the infiltration of anaesthetic solution
  The investigators ask the patients to evaluate the total pain that the infiltration of the anaesthetic solution caused using Visual Analogue Scale (VAS). The Visual Analogue Scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable.
Worst pain during the operation (VAS) | Immediately after the operation
  The investigators ask the patients to evaluate the worst pain during the operation using Visual Analogue Scale (VAS). The Visual Analogue Scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable.
Duration of anaesthesia | Postoperatively during the first 72 hours after the operation
  The investigators assess the length of the anaesthesia by asking the patients to fill an online form when they first time feel pain in the operation field or have to use pain killers.
Self-reported symptom severity and functional status | Before and 3 months postoperatively
  The investigators ask the patients to evaluate their symptoms using Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) score. It consists of the Symptom Severity Scale (SSS) containing 11 questions, and it uses a five-point Likert rating scale from 1 (no symptoms) to 5 (most severe symptoms), and Functional Status Scale (FSS), which has 8 questions assessing the degree of complaints on a five-point Likert scale from 1 (no symptoms) to 5 (most severe symptoms). Mean sum scores of both scales are calculated and used for analysis.
Patient satisfaction | 3 months postoperatively
  Patients evaluate how likely they would recommend the procedure to a fellow man using Net Promoter Score (NPS). Net Promoter Score is a measurement taken from asking patients how likely they are to recommend the procedure to others on a scale of 0-10. The higher score the better outcome.
Adverse events (AE) | 3 months postoperatively
  Health care professional assessment
Expected pain (VAS) | Before the infiltration of the anaesthetic solution
  The investigators ask the patient to evaluate the pain during the infiltration of the anaestetic solution using Visual Analogue Scale (VAS). The Visual Analogue Scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable.
Amount of perceived needle stings | Immediately after the infiltration of anaesthetic solution
  The investigators ask the patient to report how many needle stings they felt when the anaesthesia was performed.
Consumption of pain killers | Postoperatively during the first 72 hours after the operation
  The investigators record the consumption of pain killers after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yrjänä Nietosvaara, Prof., Study Director — Kuopio University Hospital
Locations (1):
- Kuopio University hospital, Department of Orthopaedics, Traumatology and Hand Surgery, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: Yes
This trial will share data with researchers who submit a methodologically sound proposal after its completion, as well as with reviewers of the journal where the trial results will be published, if necessary.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available for 15 years after the study has ended.
Access Criteria: Request must come from an EU/ETA country. The investigators do not share data outside these countries.

REFERENCES:
- [Background] Shi Q, MacDermid JC. Is surgical intervention more effective than non-surgical treatment for carpal tunnel syndrome? A systematic review. J Orthop Surg Res. 2011 Apr 11;6:17. doi: 10.1186/1749-799X-6-17. PMID 21477381
- [Background] Piazzini DB, Aprile I, Ferrara PE, Bertolini C, Tonali P, Maggi L, Rabini A, Piantelli S, Padua L. A systematic review of conservative treatment of carpal tunnel syndrome. Clin Rehabil. 2007 Apr;21(4):299-314. doi: 10.1177/0269215507077294. PMID 17613571
- [Background] Keir PJ, Rempel DM. Pathomechanics of peripheral nerve loading. Evidence in carpal tunnel syndrome. J Hand Ther. 2005 Apr-Jun;18(2):259-69. doi: 10.1197/j.jht.2005.02.001. PMID 15891983
- [Background] Kozak A, Schedlbauer G, Wirth T, Euler U, Westermann C, Nienhaus A. Association between work-related biomechanical risk factors and the occurrence of carpal tunnel syndrome: an overview of systematic reviews and a meta-analysis of current research. BMC Musculoskelet Disord. 2015 Sep 1;16:231. doi: 10.1186/s12891-015-0685-0. PMID 26323649
- [Background] Padua L, Di Pasquale A, Pazzaglia C, Liotta GA, Librante A, Mondelli M. Systematic review of pregnancy-related carpal tunnel syndrome. Muscle Nerve. 2010 Nov;42(5):697-702. doi: 10.1002/mus.21910. PMID 20976778
- [Background] Mondelli M, Giannini F, Giacchi M. Carpal tunnel syndrome incidence in a general population. Neurology. 2002 Jan 22;58(2):289-94. doi: 10.1212/wnl.58.2.289. PMID 11805259
- [Background] Shiri R, Pourmemari MH, Falah-Hassani K, Viikari-Juntura E. The effect of excess body mass on the risk of carpal tunnel syndrome: a meta-analysis of 58 studies. Obes Rev. 2015 Dec;16(12):1094-104. doi: 10.1111/obr.12324. Epub 2015 Sep 23. PMID 26395787
- [Background] Shiri R. Hypothyroidism and carpal tunnel syndrome: a meta-analysis. Muscle Nerve. 2014 Dec;50(6):879-83. doi: 10.1002/mus.24453. Epub 2014 Oct 30. PMID 25204641
- [Background] Pourmemari MH, Shiri R. Diabetes as a risk factor for carpal tunnel syndrome: a systematic review and meta-analysis. Diabet Med. 2016 Jan;33(1):10-6. doi: 10.1111/dme.12855. Epub 2015 Aug 18. PMID 26173490
- [Background] Chammas M, Boretto J, Burmann LM, Ramos RM, Dos Santos Neto FC, Silva JB. Carpal tunnel syndrome - Part I (anatomy, physiology, etiology and diagnosis). Rev Bras Ortop. 2014 Aug 20;49(5):429-36. doi: 10.1016/j.rboe.2014.08.001. eCollection 2014 Sep-Oct. PMID 26229841
- [Background] Genova A, Dix O, Saefan A, Thakur M, Hassan A. Carpal Tunnel Syndrome: A Review of Literature. Cureus. 2020 Mar 19;12(3):e7333. doi: 10.7759/cureus.7333. PMID 32313774
- [Background] Kim PT, Lee HJ, Kim TG, Jeon IH. Current approaches for carpal tunnel syndrome. Clin Orthop Surg. 2014 Sep;6(3):253-7. doi: 10.4055/cios.2014.6.3.253. Epub 2014 Aug 5. PMID 25177448
- [Background] Wang L. Guiding Treatment for Carpal Tunnel Syndrome. Phys Med Rehabil Clin N Am. 2018 Nov;29(4):751-760. doi: 10.1016/j.pmr.2018.06.009. Epub 2018 Sep 17. PMID 30293628
- [Background] Padua L, Coraci D, Erra C, Pazzaglia C, Paolasso I, Loreti C, Caliandro P, Hobson-Webb LD. Carpal tunnel syndrome: clinical features, diagnosis, and management. Lancet Neurol. 2016 Nov;15(12):1273-1284. doi: 10.1016/S1474-4422(16)30231-9. Epub 2016 Oct 11. PMID 27751557
- [Background] Wipperman J, Goerl K. Carpal Tunnel Syndrome: Diagnosis and Management. Am Fam Physician. 2016 Dec 15;94(12):993-999. PMID 28075090
- [Background] Delaunay L, Chelly JE. Blocks at the wrist provide effective anesthesia for carpal tunnel release. Can J Anaesth. 2001 Jul-Aug;48(7):656-60. doi: 10.1007/BF03016199. PMID 11495872
- [Background] Cranford CS, Ho JY, Kalainov DM, Hartigan BJ. Carpal tunnel syndrome. J Am Acad Orthop Surg. 2007 Sep;15(9):537-48. doi: 10.5435/00124635-200709000-00004. PMID 17761610
- [Background] Shiri R. Arthritis as a risk factor for carpal tunnel syndrome: a meta-analysis. Scand J Rheumatol. 2016 Oct;45(5):339-46. doi: 10.3109/03009742.2015.1114141. Epub 2016 Mar 29. PMID 27022991
- [Background] Ozdag Y, Hu Y, Hayes DS, Manzar S, Akoon A, Klena JC, Grandizio LC. Sensitivity and Specificity of Examination Maneuvers for Carpal Tunnel Syndrome: A Meta-Analysis. Cureus. 2023 Jul 24;15(7):e42383. doi: 10.7759/cureus.42383. eCollection 2023 Jul. PMID 37621797
- [Background] Iqbal HJ, Doorgakant A, Rehmatullah NNT, Ramavath AL, Pidikiti P, Lipscombe S. Pain and outcomes of carpal tunnel release under local anaesthetic with or without a tourniquet: a randomized controlled trial. J Hand Surg Eur Vol. 2018 Oct;43(8):808-812. doi: 10.1177/1753193418778999. Epub 2018 Jun 5. PMID 29871567
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Jarvinen TL, Sihvonen R, Bhandari M, Sprague S, Malmivaara A, Paavola M, Schunemann HJ, Guyatt GH. Blinded interpretation of study results can feasibly and effectively diminish interpretation bias. J Clin Epidemiol. 2014 Jul;67(7):769-72. doi: 10.1016/j.jclinepi.2013.11.011. Epub 2014 Feb 20. PMID 24560088
- [Background] Impact of blinding on estimated treatment effects in randomised clinical trials: meta-epidemiological study. BMJ. 2020 Feb 5;368:m358. doi: 10.1136/bmj.m358. No abstract available. PMID 32024659
- [Background] Tashjian RZ, Deloach J, Porucznik CA, Powell AP. Minimal clinically important differences (MCID) and patient acceptable symptomatic state (PASS) for visual analog scales (VAS) measuring pain in patients treated for rotator cuff disease. J Shoulder Elbow Surg. 2009 Nov-Dec;18(6):927-32. doi: 10.1016/j.jse.2009.03.021. Epub 2009 Jun 16. PMID 19535272
- [Derived] Heikkinen N, Nietosvaara Y, Reito A, Sirola J, Hytonen M, Savolainen A, Raisanen MP. Carpal tunnel release under local anesthesia with or without distal median nerve block: Double-blind randomized clinical trial. Scand J Surg. 2025 Mar;114(1):13-21. doi: 10.1177/14574969241277028. Epub 2024 Sep 19. PMID 39297416